CLINICAL TRIAL: NCT02046148
Title: A Phase II, Multicenter, Randomized, Observer-Blind, Controlled Study to Evaluate Safety and Immunogenicity of a Trivalent Group B Streptococcus Vaccine in Healthy Pregnant Women
Brief Title: Safety and Immunogenicity of a Trivalent Group B Streptococcus Vaccine in Healthy Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205235; V98_12 (Other: Novartis)
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: GBS Disease; Streptococcus Agalactiae
Keywords: Maternal vaccine; IgG; IgA; GBS; pregnant women

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GBS Group (Experimental): Healthy pregnant women, between and including 18-40 years of age, at 24 0/7 through 34 6/7 weeks of gestation, with the intent to breastfeed, who received a single dose of Group B Streptococcus (GBS) trivalent vaccine, injected intramuscularly. (Pregnant women are referred to as maternal subjects as the study period spans from pregnancy to Day 180 postpartum).
  Interventions: Biological: GBS trivalent vaccine
- Placebo Group (Active Comparator): Healthy pregnant women, between and including 18-40 years of age, at 24 0/7 through 34 6/7 weeks of gestation, with the intent to breastfeed, who received a single dose of Placebo, injected intramuscularly. (Pregnant women are referred to as maternal subjects as the study period spans from pregnancy to Day 180 postpartum).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GBS trivalent vaccine — Intramuscular injection - Liquid formulation of a vaccine containing polysaccharide capsules from serotypes Ia, Ib, and III of the Group B Streptococcus and conjugated to the Corynebacterium diphtheriae CRM197 carrier protein
  Arms: GBS Group
Biological: Placebo — Intramuscular injection - Normal saline
  Arms: Placebo Group

SUMMARY:
Evaluate the safety and immunogenicity of the trivalent group B streptococcus vaccine in healthy pregnant women. The study will also evaluate the levels of GBS serotype-specific antibodies in infants, placental transfer from the pregnant women to the infant and levels of antibodies in the breast milk.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women 18-40 years of age, inclusive and at 24 0/7 through 34 6/7 weeks gestation.
2. Individuals who intend to breastfeed for at least 90 days postpartum.
3. Individuals who have given written consent after the nature of the study has been explained according to local regulatory requirements.
4. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.
5. Individuals who can comprehend and comply with all study procedures and are available for follow-up.

Exclusion Criteria:

1. Individuals with history of illness or an ongoing illness that, in the opinion of the investigator, may pose additional risk to the subject if she participates in the study.
2. Individuals with known hypersensitivity to any component of the vaccine.
3. Individuals who received or plan to receive any licensed vaccine within 14 days before or after the study vaccine with the exception of inactivated influenza vaccine which may be administered up to 7 days before or after study vaccine.
4. Individuals with an infection requiring systemic antibiotic or antiviral treatment within 7 days prior to Study Day 1.
5. Individuals determined as high risk for serious obstetrical complication, including:

   * Gestational hypertension, as defined by American College of Obstetricians and Gynecologists guidelines (ACOG Practice Bulletin 2012)
   * Gestational diabetes which is not controlled by diet and exercise as per American College of Obstetricians and Gynecologists guidelines (ACOG Practice Bulletin 2013)
   * Pre-eclampsia or eclampsia as defined by American College of Obstetricians and Gynecologists guidelines (ACOG practice bulletin, 2002)
   * HIV infection
   * Obesity class II or greater (pre-pregnancy BMI≥35.0)
   * multiple pregnancy
6. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
7. Individuals who are not able to comprehend and to follow all required study procedures for the whole period of the study.
8. Individuals with known or suspected impairment of the immune system including known or suspected HIV infection or HIV-related disease, a history of or an active autoimmune disorder and receipt of immunosuppressive therapy.
9. Long term use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) within 30 days prior to enrollment. Use of inhaled, intranasal, or topical corticosteroids is allowed.
10. Individuals participating in any clinical trial with another investigational product during the pregnancy or intent to participate in another clinical study at any time during the conduct of this study.
11. Pregnant with a fetus with a known or suspected congenital anomaly
12. Individuals who are acting as study personnel or immediate family members (brother, sister, child, parent) or the spouse of study personnel.
13. Individuals with a fever (oral temperature ≥ 38°C/100.4 °F) within 3 days prior to intended study vaccination.
14. Individuals with a history of culture confirmed GBS case in the infant(s) previously born to her.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2016-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20751

REFERENCES:
- [Derived] Swamy GK, Metz TD, Edwards KM, Soper DE, Beigi RH, Campbell JD, Grassano L, Buffi G, Dreisbach A, Margarit I, Karsten A, Henry O, Lattanzi M, Bebia Z. Safety and immunogenicity of an investigational maternal trivalent group B streptococcus vaccine in pregnant women and their infants: Results from a randomized placebo-controlled phase II trial. Vaccine. 2020 Oct 14;38(44):6930-6940. doi: 10.1016/j.vaccine.2020.08.056. Epub 2020 Sep 1. PMID 32883555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in United States.
Period: Overall Study
Arm/Group | GBS Group | Placebo Group
Started | 49 | 26
Completed | 48 | 23
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GBS Group | Placebo Group | Total
Number analyzed (Participants) | 49 | 26 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.4 (4.2) | 29.4 (5.1) | 29.4 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 26 | 75
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Serotype Ia GBS IgG Levels in Infant Serum at Delivery and at Days 42 and 90 of Age
Description: To evaluate serotype-specific Ia GBS serum IgG antibody levels (anti-Ia) in infants born to maternal subjects receiving the GBS trivalent vaccine, as measured at birth, Day 42 and Day 90 of age. Antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL).
Time Frame: At Birth, Day 42 and Day 90
Population: All screened subjects who signed informed consent form, provided demographic data and/or baseline screening assessments, were randomized and assigned a study subject ID, who correctly received the study vaccine, who had no major protocol deviation, and who provided at least one evaluable serum sample at the relevant time points.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 44 | 23
µg/mL
  Anti-Ia Birth | 6.98 [3.09 to 16] | 0.24 [0.085 to 0.69]
  Anti-Ia Day 42: number analyzed (Participants) | 38 | 19
  Anti-Ia Day 42 | 6.18 [2.6 to 15] | 0.39 [0.12 to 1.23]
  Anti-Ia Day 90: number analyzed (Participants) | 37 | 16
  Anti-Ia Day 90 | 2.74 [1.2 to 6.28] | 0.33 [0.11 to 0.98]

2. Primary Outcome: Concentration of Serotype Ib GBS IgG Levels in Infant Serum at Delivery and at Days 42 and 90 of Age
Description: To evaluate serotype-specific Ib GBS serum IgG antibody levels (anti-Ib) in infants born to maternal subjects receiving the GBS trivalent vaccine, as measured at birth, Day 42 and Day 90 of age. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay
Time Frame: At Birth, Day 42 and Day 90
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 41 | 23
µg/mL
  Anti-Ib Birth | 4.65 [2.07 to 10] | 0.6 [0.22 to 1.68]
  Anti-Ib Day 42: number analyzed (Participants) | 35 | 19
  Anti-Ib Day 42 | 3.02 [1.29 to 7.07] | 0.63 [0.21 to 1.94]
  Anti-Ib Day 90: number analyzed (Participants) | 35 | 16
  Anti-Ib Day 90 | 1.81 [0.83 to 3.94] | 0.52 [0.19 to 1.45]

3. Primary Outcome: Concentration of Serotype III GBS IgG Levels in Infant Serum at Delivery and at Days 42 and 90 of Age
Description: To evaluate serotype-specific III GBS serum IgG antibody levels (anti-III) in infants born to maternal subjects receiving the GBS trivalent vaccine, as measured at birth, Day 42 and Day 90 of age. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Birth, Day 42 and Day 90
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 40 | 22
µg/mL
  Anti-III Birth | 7.97 [3.18 to 20] | 0.21 [0.064 to 0.67]
  Anti-III Day 42: number analyzed (Participants) | 38 | 19
  Anti-III Day 42 | 2.64 [1.06 to 6.56] | 0.25 [0.075 to 0.84]
  Anti-III Day 90: number analyzed (Participants) | 36 | 16
  Anti-III Day 90 | 2.01 [0.75 to 5.36] | 0.22 [0.06 to 0.78]

4. Primary Outcome: Concentration of Serotype Ia GBS IgG Levels in Maternal Serum at Pre-vaccination, at Study Day 31, at Delivery and at Days 42 and 90 Postpartum
Description: To evaluate serotype-specific (Ia) GBS serum IgG antibody levels (anti-Ia) in maternal subjects. Antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL).
Time Frame: At Day 1 (pre-vaccination), Day 31 (post-vaccination), Delivery, Days 42 and 90 (postpartum)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
µg/mL
  Anti-Ia Day 1 pre-vaccination | 0.49 [0.29 to 0.82] | 0.33 [0.18 to 0.62]
  Anti-Ia Day 31 post-vaccination: number analyzed (Participants) | 43 | 25
  Anti-Ia Day 31 post-vaccination | 8.99 [4.7 to 17] | 0.4 [0.18 to 0.85]
  Anti-Ia Delivery: number analyzed (Participants) | 40 | 25
  Anti-Ia Delivery | 5.37 [2.97 to 9.71] | 0.36 [0.18 to 0.71]
  Anti-Ia Day 42 postpartum: number analyzed (Participants) | 41 | 22
  Anti-Ia Day 42 postpartum | 13 [6.91 to 24] | 0.64 [0.3 to 1.4]
  Anti-Ia Day 90 postpartum: number analyzed (Participants) | 44 | 19
  Anti-Ia Day 90 postpartum | 8.38 [4.42 to 16] | 0.58 [0.25 to 1.35]

5. Primary Outcome: Concentration of Serotype Ib GBS IgG Levels in Maternal Serum at Pre-vaccination, at Study Day 31, at Delivery and at Days 42 and 90 Postpartum
Description: To evaluate serotype-specific (Ib) GBS serum IgG antibody levels (anti-Ib) in maternal subjects. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 1 (pre-vaccination), Day 31 (post-vaccination), Delivery, Days 42 and 90 (postpartum)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 47 | 26
µg/mL
  Anti-Ib Day 1 pre-vaccination | 0.34 [0.24 to 0.48] | 0.42 [0.28 to 0.63]
  Anti-Ib Day 31 post-vaccination: number analyzed (Participants) | 39 | 25
  Anti-Ib Day 31 post-vaccination | 7.32 [3.48 to 15] | 0.47 [0.2 to 1.11]
  Anti-Ib Delivery: number analyzed (Participants) | 37 | 25
  Anti-Ib Delivery | 5.59 [2.98 to 10] | 0.41 [0.2 to 0.85]
  Anti-Ib Day 42 postpartum: number analyzed (Participants) | 38 | 20
  Anti-Ib Day 42 postpartum | 8.9 [4.72 to 17] | 0.61 [0.27 to 1.38]
  Anti-Ib Day 90 postpartum: number analyzed (Participants) | 42 | 18
  Anti-Ib Day 90 postpartum | 6.15 [3.22 to 12] | 0.53 [0.22 to 1.29]

6. Primary Outcome: Concentration of Serotype III GBS IgG Levels in Maternal Serum at Pre-vaccination, at Study Day 31, at Delivery and at Days 42 and 90 Postpartum
Description: To evaluate serotype-specific (III) GBS serum IgG antibody levels (anti-III) in maternal subjects. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 1 (pre-vaccination), Day 31 (post-vaccination), Delivery, Days 42 and 90 (postpartum)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 43 | 25
µg/mL
  Anti-III Day 1 pre-vaccination | 0.31 [0.18 to 0.54] | 0.19 [0.1 to 0.34]
  Anti-III Day 31 post-vaccination: number analyzed (Participants) | 38 | 24
  Anti-III Day 31 post-vaccination | 3.61 [1.51 to 8.61] | 0.28 [0.12 to 0.69]
  Anti-III Delivery: number analyzed (Participants) | 35 | 23
  Anti-III Delivery | 4.4 [2.1 to 9.2] | 0.27 [0.13 to 0.56]
  Anti-III Day 42 postpartum: number analyzed (Participants) | 37 | 21
  Anti-III Day 42 postpartum | 3.74 [2.24 to 6.25] | 0.26 [0.13 to 0.5]
  Anti-III Day 90 postpartum: number analyzed (Participants) | 41 | 19
  Anti-III Day 90 postpartum | 4.04 [2.43 to 6.71] | 0.3 [0.15 to 0.62]

7. Primary Outcome: Ratio Relative to Pre-vaccination Levels of Maternal Serum GBS IgG Antibody Levels - Serotype Ia, as Measured at Study Day 31, at Delivery and at Days 42 and 90 Postpartum
Description: Geometric Mean Ratio relative to pre-vaccination (Day 1) of serotype-specific (Ia) GBS serum IgG antibody concentrations (anti-Ia) in maternal subjects. Antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL).
Time Frame: At Day 31 (post-vaccination), Delivery, Days 42 and 90 (postpartum)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 44 | 25
Ratio
  Anti-Ia Day 31/Day 1: number analyzed (Participants) | 43 | 25
  Anti-Ia Day 31/Day 1 | 25 [13 to 49] | 1.05 [0.49 to 2.26]
  Anti-Ia Delivery/Day 1: number analyzed (Participants) | 40 | 25
  Anti-Ia Delivery/Day 1 | 16 [8.85 to 29] | 1.03 [0.52 to 2.04]
  Anti-Ia Day 42/Day 1: number analyzed (Participants) | 41 | 22
  Anti-Ia Day 42/Day 1 | 32 [18 to 59] | 1.55 [0.71 to 3.36]
  Anti-Ia Day 90/Day 1: number analyzed (Participants) | 44 | 19
  Anti-Ia Day 90/Day 1 | 23 [12 to 43] | 1.5 [0.64 to 3.52]

8. Primary Outcome: Ratio Relative to Pre-vaccination Levels of Maternal Serum GBS IgG Antibody Levels - Serotype Ib, as Measured at Study Day 31, at Delivery and at Days 42 and 90 Postpartum
Description: Geometric Mean Ratio relative to pre-vaccination (Day 1) of serotype-specific (Ib) GBS serum IgG antibody concentrations (anti-Ib) in maternal subjects. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 31 (post-vaccination), Delivery, Days 42 and 90 (postpartum)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 41 | 25
Ratio
  Anti-Ib Day 31/Day 1: number analyzed (Participants) | 38 | 25
  Anti-Ib Day 31/Day 1 | 21 [10 to 44] | 1.39 [0.59 to 3.26]
  Anti-Ib Delivery/Day 1: number analyzed (Participants) | 36 | 25
  Anti-Ib Delivery/Day 1 | 16 [8.72 to 31] | 1.28 [0.63 to 2.6]
  Anti-Ib Day 42/Day 1: number analyzed (Participants) | 37 | 20
  Anti-Ib Day 42/Day 1 | 28 [15 to 53] | 1.9 [0.83 to 4.34]
  Anti-Ib Day 90/Day 1: number analyzed (Participants) | 41 | 18
  Anti-Ib Day 90/Day 1 | 20 [10 to 38] | 1.75 [0.71 to 4.32]

9. Primary Outcome: Ratio Relative to Pre-vaccination Levels of Maternal Serum GBS IgG Antibody Levels - Serotype III, as Measured at Study Day 31, at Delivery and at Days 42 and 90 Postpartum
Description: Geometric Mean Ratio relative to pre-vaccination (Day 1) of serotype-specific (III) GBS serum IgG antibody concentrations (anti-III) in maternal subjects. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 31 (post-vaccination), Delivery, Days 42 and 90 (postpartum)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 37 | 24
Ratio
  Anti-III Day 31/Day 1: number analyzed (Participants) | 36 | 24
  Anti-III Day 31/Day 1 | 16 [6.44 to 40] | 0.97 [0.38 to 2.46]
  Anti-III Delivery/Day 1: number analyzed (Participants) | 31 | 23
  Anti-III Delivery/Day 1 | 21 [9.38 to 45] | 0.98 [0.45 to 2.13]
  Anti-III Day 42/Day 1: number analyzed (Participants) | 34 | 21
  Anti-III Day 42/Day 1 | 16 [9.6 to 28] | 0.99 [0.49 to 1.98]
  Anti-III Day 90/Day 1: number analyzed (Participants) | 37 | 18
  Anti-III Day 90/Day 1 | 16 [9.39 to 27] | 0.98 [0.46 to 2.1]

10. Secondary Outcome: Ratio of GBS IgG Antibody Levels - Serotype Ia in Infant Serum Relative to Maternal Serum at the Time of Delivery
Description: To evaluate the relationship of serotype-specific Ia GBS IgG antibody levels (anti-Ia) in the infant serum to the GBS IgG antibody levels in the maternal serum at the time of delivery/birth. Antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL).
Time Frame: At Delivery
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 38 | 22
Ratio | 0.75 [0.63 to 0.89] | 0.86 [0.69 to 1.07]

11. Secondary Outcome: Ratio of GBS IgG Antibody Levels - Serotype Ib in Infant Serum Relative to Maternal Serum at the Time of Delivery
Description: To evaluate the relationship of serotype-specific Ib GBS IgG antibody levels (anti-Ib) in the infant serum to the GBS IgG antibody levels in the maternal serum at the time of delivery/birth. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Delivery
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 34 | 22
Ratio | 0.82 [0.73 to 0.92] | 0.95 [0.82 to 1.09]

12. Secondary Outcome: Ratio of GBS IgG Antibody Levels - Serotype III in Infant Serum Relative to Maternal Serum at the Time of Delivery
Description: To evaluate the relationship of serotype-specific III GBS IgG antibody levels (anti-III) in the infant serum to the GBS IgG antibody levels in the maternal serum at the time of delivery/birth. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Delivery
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 32 | 21
Ratio | 0.62 [0.51 to 0.76] | 0.87 [0.69 to 1.1]

13. Secondary Outcome: Percentage of Maternal Subjects With Solicited Local and Solicited Systemic Adverse Events (AEs) up to 30 Minutes
Description: Percentage and frequency of maternal subjects with solicited local and solicited systemic AEs up to Study Day 7 and calculated for four time intervals after vaccination: 30 minutes, Study Days 1-3 (without 30 min), Study Days 4-7, Study Days 1-7 (without 30 min). Threshold for Ecchymosis, Erythema, Swelling and Induration: Grade 0 (<25 mm), Any (≥ 25 mm). Systemic fever includes subjects with body temperature ≥ 38 °C irrespective of route of measurement.
Time Frame: Up to 30 minutes post-vaccination
Population: All screened subjects who signed informed consent form, provided demographic data and/or baseline screening assessments, were randomized and assigned a study subject ID and who received a study vaccination and who provided data on post-vaccination local or systemic adverse events.
Measure: Number; unit: Percentage of Maternal Subjects
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Percentage of Maternal Subjects
  Local Ecchymosis | 0 | 0
  Local Erythema | 0 | 0
  Local Induration | 0 | 0
  Local Swelling | 0 | 0
  Local Pain | 3 | 2
  Local Warmth | 0 | 0
  Systemic Arthralgia | 0 | 0
  Systemic Chills | 0 | 0
  Systemic Fatigue | 0 | 0
  Systemic Headache | 1 | 0
  Systemic Change in eating Habits | 0 | 0
  Systemic Myalgia | 1 | 0
  Systemic Nausea | 1 | 0
  Systemic Rash | 0 | 0
  Systemic Urticaria | 0 | 0
  Systemic Fever (≥ 38°C) | 0 | 0

14. Secondary Outcome: Percentage of Maternal Subjects With Solicited Local and Solicited Systemic AEs - Study Days 1-3
Description: as for outcome 13
Time Frame: During Study Days 1-3 (from 6 hours through Day 3 post-vaccination)
Population: as for outcome 13
Measure: Number; unit: Percentage of Maternal Subjects
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Percentage of Maternal Subjects
  Local Ecchymosis: number analyzed (Participants) | 48 | 25
  Local Ecchymosis | 0 | 0
  Local Erythema: number analyzed (Participants) | 48 | 25
  Local Erythema | 0 | 0
  Local Induration | 0 | 0
  Local Swelling | 0 | 0
  Local Pain | 24 | 8
  Local Warmth | 3 | 0
  Systemic Arthralgia | 1 | 2
  Systemic Chills: number analyzed (Participants) | 48 | 25
  Systemic Chills | 0 | 1
  Systemic Fatigue | 13 | 6
  Systemic Headache | 5 | 3
  Systemic Loss of appetite | 4 | 2
  Systemic Myalgia | 1 | 2
  Systemic Nausea | 7 | 2
  Systemic Rash | 1 | 0
  Systemic Urticaria | 1 | 0
  Systemic Fever (≥ 38°C) | 0 | 0

15. Secondary Outcome: Percentage of Maternal Subjects With Solicited Local and Solicited Systemic AEs - Study Days 4-7
Description: as for outcome 13
Time Frame: During Study Days 4-7
Population: as for outcome 13
Measure: Number; unit: Percentage of Maternal Subjects
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Percentage of Maternal Subjects
  Local Ecchymosis: number analyzed (Participants) | 48 | 25
  Local Ecchymosis | 0 | 0
  Local Erythema: number analyzed (Participants) | 48 | 25
  Local Erythema | 0 | 0
  Local Induration | 0 | 0
  Local Swelling | 0 | 0
  Local Pain | 5 | 1
  Local Warmth | 0 | 0
  Systemic Arthralgia | 1 | 1
  Systemic Chills: number analyzed (Participants) | 48 | 25
  Systemic Chills | 1 | 0
  Systemic Fatigue | 8 | 2
  Systemic Headache | 3 | 2
  Systemic Loss of appetite | 2 | 1
  Systemic Myalgia | 1 | 1
  Systemic Nausea | 1 | 1
  Systemic Rash | 0 | 0
  Systemic Urticaria | 0 | 0
  Systemic Fever (≥ 38°C) | 0 | 0

16. Secondary Outcome: Percentage of Maternal Subjects With Solicited Local and Solicited Systemic AEs - Study Days 1-7
Description: Percentage and frequency of maternal subjects with solicited local and solicited systemic adverse events up to Study Day 7 and calculated for four time intervals after vaccination: 30 minutes, Study Days 1-3 (without 30 min), Study Days 4-7, Study Days 1-7 (without 30 min). Threshold for Ecchymosis, Erythema, Swelling and Induration: Grade 0 (<25 mm), Any (≥ 25 mm). Systemic fever includes subjects with body temperature ≥ 38 °C irrespective of route of measurement.
Time Frame: During Study Days 1-7 (from 6 hours through Day 7 post-vaccination)
Population: as for outcome 13
Measure: Number; unit: Percentage of Maternal Subjects
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Percentage of Maternal Subjects
  Local Ecchymosis: number analyzed (Participants) | 48 | 25
  Local Ecchymosis | 0 | 0
  Local Erythema: number analyzed (Participants) | 48 | 25
  Local Erythema | 0 | 0
  Local Induration | 0 | 0
  Local Swelling | 0 | 0
  Local Pain | 24 | 8
  Local Warmth | 3 | 0
  Systemic Arthralgia | 2 | 2
  Systemic Chills: number analyzed (Participants) | 48 | 25
  Systemic Chills | 1 | 1
  Systemic Fatigue | 18 | 6
  Systemic Headache | 6 | 3
  Systemic Loss of appetite | 6 | 2
  Systemic Myalgia | 2 | 2
  Systemic Nausea | 7 | 3
  Systemic Rash | 1 | 0
  Systemic Urticaria | 1 | 0
  Systemic Fever (≥ 38°C) | 0 | 0

17. Secondary Outcome: Percentage of Maternal Subjects With Any Unsolicited AEs
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product at any dose that does not necessarily have to have a causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product. This definition includes inter-current illnesses or injuries and exacerbation of pre-existing conditions.
Time Frame: From Study Day 1 through Study Day 31
Population: All screened subjects who signed informed consent form, provided demographic data and/or baseline screening assessments, were randomized and assigned a study subject ID and who received a study vaccination and who provided data on unsolicited adverse events.
Measure: Number; unit: Percentage of Maternal Subjects
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 49 | 26
Percentage of Maternal Subjects | 18 | 6

18. Secondary Outcome: Percentage of Maternal Subjects With Serious Adverse Events (SAEs), Unsolicited Medically Attended AEs (MAEs) and Unsolicited AEs Leading to Study Withdrawal (AEs Lead. Wthwal)
Description: An SAE is defined as any untoward medical occurrence that at any dose results in one or more of the following: death; life-threatening; that does not refer to an event which hypothetically might have caused death if it were more severe; required or prolonged hospitalization; persistent or significant disability/incapacity; congenital anomaly/or birth defect; any important and significant medical event that may not be immediately life-threatening or resulting in death or hospitalization but, based upon appropriate medical judgement, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above. An MAE is defined as an adverse event that leads to an unscheduled visit to a healthcare practitioner.
Time Frame: From Study Day 1 through Study Day 31
Population: as for outcome 17
Measure: Number; unit: Percentage of Maternal Subjects
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 49 | 26
Percentage of Maternal Subjects
  Any SAE from Day 1 to Day 31 | 1 | 0
  Any MAE from Day 1 to Day 31 | 10 | 4
  Any AE lead. Wthwal Day 1 to Day 31 | 0 | 0

19. Secondary Outcome: Percentage of Maternal Subjects With SAEs, Unsolicited MAEs and Unsolicited AEs Leading to Study Withdrawal (AEs Lead. Wthwal)
Description: as for outcome 18
Time Frame: From Study Day 32 through Day 180 postpartum
Population: as for outcome 17
Measure: Number; unit: Percentage of Maternal Subjects
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 49 | 26
Percentage of Maternal Subjects
  Any SAE from Day 32 to Day 180 | 7 | 4
  Any MAE from Day 32 to Day 180 | 38 | 17
  Any AE lead. Wthwal Day 32 to Day 180 | 0 | 0

20. Secondary Outcome: Percentage of Infants With SAEs, Unsolicited MAEs and AEs Leading to Study Withdrawal
Description: as for outcome 18
Time Frame: From Birth through Day 180 of age
Population: Infants born to screened subjects who signed informed consent form, provided demographic data and/or baseline screening assessments, were randomized and assigned a study subject ID and who received a study vaccination and who provided data on unsolicited adverse events.
Measure: Number; unit: Percentage of Infant Subjects
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Percentage of Infant Subjects
  Any SAE | 7 | 3
  Any MAE | 34 | 15
  Any AE lead. Wthwal | 0 | 0

21. Secondary Outcome: Birth Weight of Infants (Mean-Standard Deviation)
Description: Weight at birth was summarized by reporting the mean and standard deviation,
Time Frame: At Birth
Population: Infants born to screened subjects who signed informed consent form, provided demographic data and/or baseline screening assessments, were randomized and assigned a study subject ID and who received a study vaccination.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Kilogram | 3.44 (0.45) | 3.32 (0.40)

22. Secondary Outcome: Birth Weight of Infants (Median, Minimum and Maximum)
Description: Weight at birth was summarized by reporting the median and the minimum and maximum.
Time Frame: At Birth
Population: as for outcome 21
Measure: Median (Full Range); unit: Kilogram
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Kilogram | 3.5 [2.3 to 4.5] | 3.3 [2.7 to 4.4]

23. Secondary Outcome: Birth Length and Head Circumference of Infants (Mean - Standard Deviation)
Description: Length and head circumference at birth were summarized by reporting the mean and standard deviation.
Time Frame: At Birth
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 46 | 25
Centimeter
  Lenght mean | 51.35 (2.26) | 49.70 (2.17)
  Head circumference mean | 34.4 (1.51) | 34.48 (1.08)

24. Secondary Outcome: Birth Length and Head Circumference of Infants (Median - Minimum and Maximum)
Description: Length and head circumference at birth were summarized by reporting the median and minimum and maximum
Time Frame: At birth
Population: as for outcome 21
Measure: Median (Full Range); unit: Centimeter
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 46 | 25
Centimeter
  Lengh Median | 52.0 [45.0 to 56.0] | 50.0 [45.7 to 55.0]
  Head circumference Median | 35.0 [32.0 to 37.0] | 34.0 [33.0 to 37.0]

25. Secondary Outcome: Infants Apgar Scores (Mean - Standard Deviation)
Description: Apgar (Appearance, Pulse, Grimace response, Activity and Respiration) test to evaluate the new-born's physical condition. Apgar score between 0 and 10 (highest score possible). If 1 and 5 minutes Apgar score were normal, 10 minutes Apgar score might not be required.
Time Frame: At 1, 5 and 10 minutes
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Scores on a scale
  Mean 1 minute | 8.13 (1.16) | 8.23 (0.51)
  Mean 5 minutes: number analyzed (Participants) | 47 | 26
  Mean 5 minutes | 8.89 (0.48) | 8.88 (0.43)
  Mean 10 minutes: number analyzed (Participants) | 2 | 1
  Mean 10 minutes | 8.5 (0.71) | 9.0 (NA) — Standard Deviation indeterminated (denominator =0)

26. Secondary Outcome: Infants Apgar Scores (Median, Minimum and Maximum)
Description: Apgar (Appearance, Pulse, Grimace response, Activity and Respiration) test to evaluate the new-born's physical condition. Apgar scores between 0 and 10 (highest score possible). If 1 and 5 minutes Apgar score were normal, 10 minutes Apgar score might not be required.
Time Frame: At 1, 5 and 10 minutes
Population: as for outcome 21
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 26
Scores on a scale
  Median 1 minute | 8.0 [1.0 to 9.0] | 8.0 [7.0 to 9.0]
  Median 5 minutes: number analyzed (Participants) | 47 | 26
  Median 5 minutes | 9.0 [7.0 to 10] | 9.0 [8.0 to 10]
  Median 10 minutes: number analyzed (Participants) | 2 | 1
  Median 10 minutes | 8.5 [8.0 to 9.0] | 9.0 [9.0 to 9.0]

27. Secondary Outcome: Descriptive Statistics for the Score for the Long-term Developmental Outcome Assessed by Bayley Scales of Infant and Toddler Development 3rd Edition Screening Test (PsychCorp) in Infants (Mean - Standard Deviation)
Description: Long-term developmental outcome assessed by Bayley Scales of Infant and Toddler Development 3rd edition Screening Test (PsychCorp). The screening test measured three domains: cognitive, language (receptive vs expressive communication), and motor (fine vs gross). Scaled scores range from 1 to 19 with a mean of 10 and a standard deviation of 3. The scores were summarized by reporting the mean and standard deviation.
Time Frame: At Day 180 of age
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 23
Scores on a scale
  Cognitive mean | 11.2 (1.7) | 11.7 (2.0)
  Receptive Communication mean | 8.8 (2.0) | 9.8 (2.5)
  Expressive Communication mean | 8.4 (2.0) | 8.9 (2.0)
  Fine Motor mean | 9.0 (1.5) | 9.5 (1.5)
  Gross Motor mean | 9.8 (1.9) | 10.3 (2.0)

28. Secondary Outcome: Descriptive Statistics for the Score for the Long-term Developmental Outcome Assessed by Bayley Scales of Infant and Toddler Development 3rd Edition Screening Test (PsychCorp) in Infants (Median, Minimum and Maximum)
Description: Long-term developmental outcome assessed by Bayley Scales of Infant and Toddler Development 3rd edition Screening Test (PsychCorp). The screening test measured three domains: cognitive, language (receptive vs expressive communication), and motor (fine vs gross). Scaled scores range from 1 to 19 with a mean of 10 and a standard deviation of 3. The scores were summarized by reporting the median, minimum and maximum.
Time Frame: At Day 180 of age
Population: as for outcome 21
Measure: Median (Full Range); unit: Sores on a scale
Arm/Group | GBS Group | Placebo Group
Number analyzed (Participants) | 48 | 23
Sores on a scale
  Cognitive median | 11.0 [7 to 15] | 12.0 [8 to 16]
  Receptive Communication median | 8.0 [5 to 12] | 9.0 [6 to 14]
  Expressive Communication median | 8.5 [5 to 13] | 9.0 [5 to 11]
  Fine Motor median | 9.0 [6 to 12] | 10.0 [7 to 13]
  Gross Motor median | 10.0 [3 to 15] | 11.0 [7 to 14]

ADVERSE EVENTS:
Time Frame: Solicited and Unsolicited AEs within the 31-day post-vaccination period for maternal subjects; SAEs from Study Day 1 to Day 180 postpartum for maternal subjects and from Birth up to Day 180 of age for Infants.
Arm/Group | GBS Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/26
Serious Adverse Events (participants affected / at risk) | 8/49 | 4/26
Other Adverse Events (participants affected / at risk) | 45/49 | 18/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | GBS Group (N=49) | Placebo Group (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Maternal subjects
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Maternal subjects
Amniotic cavity infection (Infections and infestations) | 1 (1) | 0 (0) — Maternal subjects
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0) — Maternal subjects
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Maternal subjects
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Maternal subjects
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (2) — Maternal subjects
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Maternal subjects
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Maternal subjects
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Maternal subjects
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) — Maternal subjects
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1/48 (1) | 1 (1) — Infant subjects
Polydactyly (Congenital, familial and genetic disorders) | 1/48 (1) | 0 (0) — Infant subjects
Hyperbilirubinaemia (Hepatobiliary disorders) | 1/48 (1) | 1 (1) — Infant subjects
Bronchiolitis (Infections and infestations) | 1/48 (1) | 0 (0) — Infant subjects
Parainfluenzae virus infection (Infections and infestations) | 1/48 (1) | 0 (0) — Infant subjects
Urinary tract infection (Infections and infestations) | 0/48 (0) | 1 (1) — Infant subjects
Hypoglycaemia (Metabolism and nutrition disorders) | 1/48 (1) | 0 (0) — Infant subjects
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 1/48 (1) | 0 (0) — Infant subjects
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBS Group (N=49) | Placebo Group (N=26)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 10 (11) | 4 (4)
FATIGUE (General disorders) | 18 (21) | 6 (7)
INJECTION SITE ERYTHEMA (General disorders) | 11 (13) | 5 (5)
INJECTION SITE HAEMORRHAGE (General disorders) | 2 (2) | 2 (2)
INJECTION SITE INDURATION (General disorders) | 5 (6) | 2 (2)
INJECTION SITE PAIN (General disorders) | 25 (26) | 8 (8)
INJECTION SITE SWELLING (General disorders) | 1 (1) | 3 (3)
INJECTION SITE WARMTH (General disorders) | 3 (3) | 0 (0)
MASTITIS (Infections and infestations) | 3 (3) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 2 (3) | 2 (2)
SINUSITIS (Infections and infestations) | 3 (3) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (6) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 1 (1)
PERINEAL INJURY (Injury, poisoning and procedural complications) | 10 (10) | 5 (5)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
HEADACHE (Nervous system disorders) | 8 (11) | 5 (6)
GESTATIONAL HYPERTENSION (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
OLIGOHYDRAMNIOS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
POSTPARTUM HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.